CLINICAL TRIAL: NCT05261581
Title: Evaluation of Erector Spina Plane Block(ESPB)'s Effectiveness on Patients With Lumbar Radiculopathy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficulties about the method of the study
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13.01.2022-E.46715-23/1
Record Dates: First submitted 2022-02-02; First posted 2022-03-02 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Radiculopathy; Radiculopathy Lumbar; Pain, Back
MeSH Terms: conditions — Radiculopathy; Back Pain | interventions — Anti-Inflammatory Agents, Non-Steroidal; Anti-Inflammatory Agents; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients that will get ESPB, NSAID and exercise programme
  Interventions: Procedure: Erector Spinae Plane Block; Drug: NSAID; Behavioral: Home Exercise Programme
- Control (Active Comparator): Patients that will only get NSAID and exercise programme
  Interventions: Drug: NSAID; Behavioral: Home Exercise Programme

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector spinae block (ESB) is an ultrasound-guided interfascial plane block. The local anesthetic is injected using ultrasound guidance superficial to transverse process and deep to erector spinae muscle group
  Arms: Intervention
Drug: NSAID — Non-steroidal anti-inflammatory drugs (NSAIDs) are medicines that are widely used to relieve pain, reduce inflammation.
  Other Names: Anti-inflammatory/Analgesic Treatment
Behavioral: Home Exercise Programme — Home exercise programme will include some stretches that aid in pain relief by helping take stress off the low back and hips, core stabilization exercises and postural exercises.
  Other Names: Exercise

SUMMARY:
A new regional anaesthetic block technique is described in this issue of Anaesthesia by Chin et al. whereby local anaesthetic is injected within a plane beneath the erector spinae muscle to achieve analgesia for abdominal surgery. After this the block has been used successfully for many implications such as post-herpetic neuralgia, thoracic and abdominal chronic or acute pain management, rib fractures, breast surgery, chronic cancer pain and etc. Cadaveric and radiologic data showed that contrast injected into the tissue plane deep to erector spinae muscle and superficial to the transverse processes and intertransverse connective tissues penetrates anteriorly to anesthetize the spinal nerves. And some cadeveric studies resulted with where both the dorsal and ventral rami of the thoracic spinal nerves were marked with dye after ESPB. Some studies even showed that dye reached to the epidural space. In this manner we we hypothesize that ESPB could be effective with radiculopathy pain.

DETAILED DESCRIPTION:
Forero et al. proposed in 2016 an interfascial block to provide analgesia to patients suffering from thoracic chronic pain consisting of an injection of local anesthetic inside the erector spinae plane (ESP). As stated by the authors in their original work, the discovery of this technique was casual, but subsequent observations showed that this "casual" technique had a wide range of possible indications not only to thoracic area but varying from chronic to acute traumatic pain, from thoracic to orthopedic surgery, from children to elderly patients.

There are three groups of muscles involved in this block: erector spinae muscles group, transverso-spinal muscles group and levatores rostrum. Erector spinae muscles are not a single muscle, but a really complex muscular group formed by ileocostalis muscles, longissimus muscles and spinalis muscles. These muscles link bone components of the back to each other: the spinous process to spinous process, rib to rib and transverse process to transverse process.Deep to this group of muscles, we find the transverso-spinal group of muscles connecting the transverse processes to the spinous processes (semispinalis, multifidus, rotatores), and deeper still are the levatores rostrum, originating from the transverse processes and inserting into the ribs. Together, all these muscles act as a geometrical structure that would facilitate the spread of local anesthetic.

The ESP block's therapeutic effect is attributed to the cranial-caudal spread of local anesthetic over multiple vertebral levels in the musculofascial plane deep to the erector spinae muscle, accompanied by diffusion anteriorly into the contiguous paravertebral and intercostal spaces, where the local anesthetic then acts on the ventral and dorsal rami of spinal nerves. The subsequent realization that the erector spinae muscle extends from the lumbar spine to cervical spine led to extrapolation of the ESP block for many different indications in different regions of the body.

Since after Forero's proposition in 2016 many researchers successfully tried ESPB primarily in post-operative pain and acute trauma pain management. More recently there have been some studies focusing on musculoskeletal originated pain such as myofascial pain syndrome, chronic shoulder pain/frozen shoulder etc. In this manner we hypothesize that ESPB could be effective for reducing pain effectively in a short treatment time. And considering other spinal interventions for radiculopathy pain such as transforaminal/epidural blocks require more skilled stuff, scopy device and a special place for it. Since ESPB can be done via ultrasonography and needs less stuff we also think that it can be a more cost efficient treatment choice for radiculopathy pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75
* MRI proven radiculopathy
* Pain level on NRS should be at least 4 and above

Exclusion Criteria:

* Congenital or acquired musculospinal deformities
* Pregnancy or lactation
* Systemic inflammatory or infectious diseases
* Patients with high risk of bleeding(usage of coumadin etc)
* Malignancy
* Neuromuscular diseases
* Unstable psychiatric condition
* Patient get any kind of intervention(transforaminal or epidural injections, radiofrequency treatment etc) to the pain source

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain Assesment | Change from Baseline NPRS at 1st and 3rd months
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).Numerical Rating Scales have shown high correlations with other pain-assessment tools in several studies. The feasibility of its use and good compliance have also been proven.
The Health Assessment Questionnaire (HAQ) | Change from Baseline HAQ at 1st and 3rd months
  The HAQ was developed as a comprehensive measure of outcome in patients with a wide variety of rheumatic diseases. It has also been applied to patients with man diseases and in studies of normal aging. It should be considered a generic rather than a disease-specific instrument. Its focus is on self-reported patient-oriented outcome measures, rather than process measures.
  The Aides and Devices are assigned to the specific 8 HAQ sections as follows:
  Dressing: Devices used for dressing (button hook, zipper pull, shoe horn, etc.) Arising: Special or built up chair Eating: Built up or special utensils Walking: Cane, Walker, Crutches, Wheelchair Hygiene: Bathtub bar, Long-handled appliances in bathroom, Raised toilet seat Reach: Long-handled appliances for reach Grip: Jar opener for jars previously opened Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section.
Oswestry Low Back Pain Disability Questionnaire | Change from Baseline ODI at 1st and 3rd months
  The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain.The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel.
  Each topic category is followed by 6 statements describing different potential scenarios in the patient's life and the patient checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Roland-Morris Disability Questionnaire | Change from Baseline RMQ at 1st and 3rd months
  RMQ is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. The RMQ has been shown to yield reliable measurements, which are valid for inferring the level of disability, and to be sensitive to change over time for groups of patients with low back pain. A patient taking the survey agrees or disagrees with these statements (Yes/No).
  The final score, out of 24 represents the degree of disability due to low back pain. A maximum score of 24 indicates the greatest degree of disability from back pain. This score may be used to monitor the pain and symptoms of patients with back pain over time.

SECONDARY OUTCOMES:
Change in Lomber Range of Motion(ROM) | Change from Baseline Lomber ROM at 1st and 3rd months
  The Lumbar Spine normal active range of motion is as follows:
  Flexion: 70-90* Extension: 30* Lateral Flexion: 30* Rotation: 30* Decreased in Range of motion in lumbar spine mostly caused by muscle/fascia adhesion and tightness limiting your mobility. Another more likely scenario is that fixation in vertebra or another cause of pain. The motion restriction and muscle tightness often exist together but can be separate as well.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Forero M, Rajarathinam M, Adhikary SD, Chin KJ. Erector spinae plane block for the management of chronic shoulder pain: a case report. Can J Anaesth. 2018 Mar;65(3):288-293. doi: 10.1007/s12630-017-1010-1. Epub 2017 Nov 13. PMID 29134518
- [Background] Sotome S, Sawada A, Wada A, Shima H, Kutomi G, Yamakage M. Erector spinae plane block versus retrolaminar block for postoperative analgesia after breast surgery: a randomized controlled trial. J Anesth. 2021 Feb;35(1):27-34. doi: 10.1007/s00540-020-02855-y. Epub 2020 Sep 11. PMID 32915300
- [Background] Ivanusic J, Konishi Y, Barrington MJ. A Cadaveric Study Investigating the Mechanism of Action of Erector Spinae Blockade. Reg Anesth Pain Med. 2018 Aug;43(6):567-571. doi: 10.1097/AAP.0000000000000789. PMID 29746445
- [Background] Tulgar S, Selvi O, Senturk O, Serifsoy TE, Thomas DT. Ultrasound-guided Erector Spinae Plane Block: Indications, Complications, and Effects on Acute and Chronic Pain Based on a Single-center Experience. Cureus. 2019 Jan 2;11(1):e3815. doi: 10.7759/cureus.3815. PMID 30868029
- [Background] Tulgar S, Thomas DT, Suslu H. Ultrasound guided erector spinae plane block relieves lower cervical and interscapular myofascial pain, a new indication. J Clin Anesth. 2019 Mar;53:74. doi: 10.1016/j.jclinane.2018.10.008. Epub 2018 Oct 19. No abstract available. PMID 30343227
- [Background] De Cassai A, Bonvicini D, Correale C, Sandei L, Tulgar S, Tonetti T. Erector spinae plane block: a systematic qualitative review. Minerva Anestesiol. 2019 Mar;85(3):308-319. doi: 10.23736/S0375-9393.18.13341-4. Epub 2019 Jan 4. PMID 30621377
- [Background] Takahashi H, Suzuki T. Erector spinae plane block for low back pain in failed back surgery syndrome: a case report. JA Clin Rep. 2018 Aug 27;4(1):60. doi: 10.1186/s40981-018-0198-6. PMID 32026979
- [Background] Tulgar S, Balaban O. Spread of local anesthetic in erector spine plane block at thoracic and lumbar levels. Reg Anesth Pain Med. 2019 Jan;44(1):134-135. doi: 10.1136/rapm-2018-000027. No abstract available. PMID 30640667